CLINICAL TRIAL: NCT02056197
Title: Influence of an Exercise Program for Trunk Stabilization Performed in Stable and Unstable Surfaces for Chronic Low Back Pain: Single-blind, Randomized Controlled Clinical Trial.
Brief Title: Influence of an Exercise for Trunk Stabilization Performed in Stable and Unstable Surfaces for Chronic Low Back Pain.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Paulo Roberto Garcia Lucareli, Professor, University of Nove de Julho
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: PL002
Record Dates: First submitted 2014-01-28; First posted 2014-02-05 (Estimated); Last update posted 2014-02-05 (Estimated); Status verified 2014-01

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Shortwave 30 minutes.
  Interventions: Other: Placebo
- Stable (Active Comparator): Stable surface exercises
  Interventions: Other: Stable surface exercises
- Unstable (Experimental): Unstable surface exercises
  Interventions: Other: Unstable surface exercises

INTERVENTIONS:
Other: Placebo — Shortwave
  Arms: Placebo
Other: Stable surface exercises — Stable surface exercises
  Arms: Stable
Other: Unstable surface exercises
  Arms: Unstable

SUMMARY:
Motor control exercises have demonstrated a good option for recovery from chronic low back pain. The purpose of this study is investigated the effectiveness of an exercise program for trunk stabilization performed in stable and unstable surfaces for people with nonspecific chronic low back pain (NCLBP). Patients will be randomly divided into 3 groups; control group will receive placebo treatment with shortwave; stable group will receive an exercise protocol to stabilize the trunk on a stable surface and unstable group will receive the same exercise protocol but performed on an unstable surface.

We hypothesized the unstable group will present pain reduction and functional improvement.

ELIGIBILITY:
Inclusion Criteria:

* Non-specific low back pain
* Sedentary
* Previous low back pain last 6 months

Exclusion Criteria:

* Traumatic, inflammatory, infectious or tumours etiology
* Positive neurological findings (leg pain)
* Pregnancy
* Previous spine or lower limb surgery
* Contraindicated for short-waves aplication

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-05; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Pain Scores on the Visual Analog Scale | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Paulo RG Lucareli, PhD, Study Chair — University of Nove de Julho
Locations (1):
- Universidade Nove de Julho, São Paulo, São Paulo, Brazil